CLINICAL TRIAL: NCT00086827
Title: A Phase II Study of Single Agent Depsipeptide (FK228) (NSC 630176; IND 51,810) in Relapsed Small Cell Lung Cancer
Brief Title: Romidepsin in Treating Patients With Relapsed Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02785; NCI-2012-02785 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CALGB-30304 (Other: Cancer and Leukemia Group B); CALGB-30304 (Other: CTEP); P30CA014236 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — romidepsin

ARMS (1):
- Treatment (romidepsin) (Experimental): Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity. Patients who have continuing tumor response or stable disease after 6 courses receive 2 additional courses beyond best response.
  Interventions: Drug: romidepsin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well FR901228 works in treating patients with recurrent small cell lung cancer. FR901228 may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response rate of patients with histologically or cytologically proven small cell lung cancer (SCLC) treated with depsipeptide in the "sensitive" relapse setting.

SECONDARY OBJECTIVES:

I. To describe the overall survival and failure-free survival of patients with histologically proven recurrent SCLC treated with depsipeptide.

II. To evaluate the toxicity of depsipeptide in patients with relapsed SCLC. III. To evaluate surrogate biological markers from peripheral blood mononuclear cells and buccal epithelial cells: p53 acetylation, histone acetylation, p21CIP1 expression.

OUTLINE:

Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity. Patients who have continuing tumor response or stable disease after 6 courses receive 2 additional courses beyond best response.

Patients are followed every 3 months for 1 year and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Either histologic or cytologic documentation of recurrent small cell lung carcinoma (SCLC)
* No more than 1 prior chemotherapy regimen; must have recurrent disease after treatment with a platinum agent (either cisplatin or carboplatin); prior chemotherapy must have been completed ≥90 days prior to documentation of relapse
* >= 4 weeks since prior radiation therapy; prior radiation therapy is allowed either in the context of curative intent combined modality treatment for limited stage disease, prophylactic cranial radiation or palliative radiation (to the chest, brain, or other sites) initially or at relapse
* Prior surgery is allowed provided patients have completely recovered from effects of procedure and >= 2 weeks have elapsed
* No prior treatment with depsipeptide
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to depsipeptide
* No current treatment with any other investigational agent or drugs known to have HDI activity (HDAC or histone deacetylase inhibitor) such as sodium valproate
* Patients with treated/controlled brain mets (defined as no need for further radiation and no requirements for steroids to control peri-tumoral edema) are eligible for this study; however, patients requiring treatment with enzyme inducing anti-convulsant drugs are not eligible; these include, but are not limited to, phenytoin, phenobarbital, carbamazepine, felbamate and primidone
* All Patients must have Measurable Disease

  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension; the longest diameter of measurable lesions must be >= 20 mm with conventional techniques or >= 10 mm with spiral CT scan; lesions that are not considered measurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
    * Tumor lesions situated in a previously irradiated area
* ECOG Performance Status 0-1
* No significant cardiac disease, including:
* Congestive heart failure that meets New York Heart Association (NYHA) class III/IV definitions, history of myocardial infarction within one year of study entry, uncontrolled dysrhythmias, or poorly controlled angina
* History of serious ventricular arrhythmia (VT or VF, >= 3 beats in a row), QTc >= 500 msec, or LVEF =< 40% by MUGA
* Evidence of left ventricular hypertrophy by echocardiographic criteria or by EKG criteria (Cornell voltage criteria):

For Men: S in V3 plus R in aVL > 2.8 mV (28mm) For Women: S in V3 + R in aVL > 2.0 mV (20mm)

* Patients may not be co-medicated with an agent that causes QTc prolongation
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, HIV-positive patients receiving combination anti-retroviral therapy are not eligible because of possible pharmacokinetic interactions with depsipeptide
* No current treatment with potassium wasting diuretics (e.g., hydroclorothiazide); patients on such diuretics should be switched to a potassium sparing diuretic or another antihypertensive medication prior to registration
* Granulocytes >= 1,500/μl
* Platelets >= 100,000/μl
* Total Bilirubin =< 1.5 x ULN
* AST (SGOT) =< 2.5 x ULN
* Creatinine ≤1.5 x ULN OR Calculated Creatinine Clearance >= 60 ml/min

Exclusion Criteria:

* Non-pregnant and non-nursing because of significant risk to the fetus/infant; the effects of depsipeptide on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because histone deacetylase inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to and for the entire duration of participation and for at least 6 weeks after completion of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-05; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Up to 4 years
  95% confidence intervals will be estimated.

SECONDARY OUTCOMES:
Overall survival | Between registration and death, assessed up to 4 years
  Described using Kaplan-Meier curves.
Failure-free survival | The time between registration and disease progression or death, assessed up to 4 years
  Described using Kaplan-Meier curves.
The frequency of toxicity occurrence, graded using the NCI CTCAE version 3.0 | Up to 4 years
  Tabulated by type and grade.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Otterson, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Ohio State University, Columbus, Ohio, United States